CLINICAL TRIAL: NCT06036277
Title: Influence of Immersion in Water During Labor on the Request of Epidural Anesthesia by Pregnant Women in Case of a Desire for Physiological Delivery
Brief Title: Influence of Immersion in Water During Labor on the Request of Epidural Anesthesia by Pregnant Women
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN702023/CHUSTE
Record Dates: First submitted 2023-08-21; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-07

CONDITIONS: Delivery; Labor Pain
Keywords: Water immersion; Waterbirth; Childbirth; Labor pain; Epidural anesthesia; Physiological delivery; Pregnant women; General medicine
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Women who wish to give birth without epidural anesthesia and have benefited of water immersion during labor
  Interventions: Other: General data; Other: Other data
- Control group: Women who wish to give birth without epidural anesthesia and have not benefited of water immersion during labor
  Interventions: Other: General data; Other: Other data

INTERVENTIONS:
Other: General data — General data will be collected to ensure that both groups are comparable : maternal age, maternal BMI, gestational age, parity, number of children in current pregnancy, history of caesarian section, newborn child weight
Other: Other data — Other data collected will be used to estimate primary and secondary outcomes : request for an epidural anesthesia by the parturient, medical indication for peridural anesthesia, duration of childbirth, delivery methods, occurrence of maternal or neonatal complications.

SUMMARY:
Women are showing a growing interest in less medicalized childbirth. According to the french 2021 perinatal survey, 52.2% of women want to limit medical procedures and 38.2% of women want childbirth without epidural anesthesia. Between 77 and 82% of deliveries nevertheless lead to an epidural anesthesia. The painful feeling seems to be the main motivation for using this mode of anesthesia.

DETAILED DESCRIPTION:
In the scientific literature, few data from clinical studies focus on the effects of immersion in water during childbirth. The analgesic effects of immersion in water to lessen the painful experience are yet to be proven. The opening of a physiological delivery room with a bathtub at the Saint-Etienne University Hospital since October 2020 provides data that has not been exploited yet and could make possible to answer the question of the analgesic effects of immersion in water during labour. The difficulties of analysis and the subjectivity of the painful feeling led us to consider the request of epidural anesthesia as the main analysis criterion.

ELIGIBILITY:
Inclusion Criteria:

* All women who used the physiological delivery room of the Saint-Etienne University Hospital between October 2020 and December 2022.

Exclusion Criteria:

* Absence of physiological desire for childbirth.
* Medical indication for epidural anesthesia.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnent women who used the physiological delivery room of the Saint-Etienne University Hospital between October 2020 and December 2022.
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of requests for epidural anesthesia by parturients | Day 0
  Retrospective collection of medical data from the computer software Easily in Saint-Etienne university hospital center.

SECONDARY OUTCOMES:
Duration of the first stage of childbirth | Day 0
  Retrospective collection of medical data from the computer software Easily in Saint-Etienne university hospital center.
Duration of the second stage of childbirth | Day 0
  Retrospective collection of medical data from the computer software Easily in Saint-Etienne university hospital center.
Duration of the third stage of childbirth | Day 0
  Retrospective collection of medical data from the computer software Easily in Saint-Etienne university hospital center.
Number of instrumental extractions | Day 0
  Retrospective collection of medical data from the computer software Easily in Saint-Etienne university hospital center.
Number of caesareans | Day 0
  Retrospective collection of medical data from the computer software Easily in Saint-Etienne university hospital center.
Number and degree of perineal tear | Day 0
  Retrospective collection of medical data from the computer software Easily in Saint-Etienne university hospital center.
Use of episiotomy by the obstetrical team | Day 0
  Retrospective collection of medical data from the computer software Easily in Saint-Etienne university hospital center.
Estimated postpartum hemorrhagic volume and occurrence of postpartum hemorrhage | Day 0
  Retrospective collection of medical data from the computer software Easily in Saint-Etienne university hospital center.
Apgar score (Appearance, Pulse, Grimace, Activity, Respiration) from 0 to 10 of the child at birth | Day 0
  Retrospective collection of medical data from the computer software Easily in Saint-Etienne university hospital center.
  At 5 minutes a score of 7 to 10 is considered normal; a score of 4 to 6 is intermediate and a score of 0 to 3 is low.
Arterial pH measured at the umbilical cord | Day 0
  Retrospective collection of medical data from the computer software Easily in Saint-Etienne university hospital center.
Number of neonatal resuscitation | Day 0
  Retrospective collection of medical data from the computer software Easily in Saint-Etienne university hospital center.

CONTACTS AND LOCATIONS:
Overall Officials: Tiphaine BARJAT, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No